CLINICAL TRIAL: NCT03353662
Title: The Assessment of Sub-Regional Micronutrient Deficiencies in Ethiopia to Target Bio Fortification.
Brief Title: Sub Regional Micronutrient Survey in Ethiopia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: HarvestPlus (Other); Addis Ababa University (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Professor and Head of Human Nutrition Laboratory, Institute of Food, Nutrition and Health, ETH Zurich, Swiss Federal Institute of Technology
Other Study IDs: Ethiopia_SRMNS
Record Dates: First submitted 2017-11-13; First posted 2017-11-27 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Iron-deficiency; Vitamin A Deficiency; Zinc Deficiency
Keywords: bio fortification
MeSH Terms: conditions — Anemia, Iron-Deficiency; Vitamin A Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood Plasma will be retained, however, will only be used to measure micronutrient status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Women of Gamo Gofa: The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the women of Gamo Gofa between 15-49 years
  Interventions: Other: Women of Gamo Gofa
- Children of Gamo Gofa: The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the children of Gamo Gofa between 6 - 59 months
  Interventions: Other: Children of Gamo Gofa
- Women of West Gojjam: The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the women of West Gojjam between 15-49 years
  Interventions: Other: Women of West Gojjam
- Children of West Gojjam: The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the children of West Gojjam between 6 - 59 months
  Interventions: Other: Children of West Gojjam
- Women of Kamashi: The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the women of Kamashi between 15-49 years
  Interventions: Other: Women of Kamashi
- Children of Kamashi: The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the children of Kamashi between 6 - 59 months
  Interventions: Other: Children of Kamashi

INTERVENTIONS:
Other: Women of Gamo Gofa — The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the women of Gamo Gofa between 15-49 years by measuring hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), C-reactive protocol (CRP), alpha-1-acid glycoprotein (AGP), plasma Zn (PZn), plasma retinol and retinol binding protein (RBP), respectively.
  Groups: Women of Gamo Gofa
Other: Children of Gamo Gofa — The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the children of Gamo Gofa between 6-59 months by measuring hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), C-reactive protocol (CRP), alpha-1-acid glycoprotein (AGP), plasma Zn (PZn), plasma retinol and retinol binding protein (RBP), respectively.
  Groups: Children of Gamo Gofa
Other: Women of West Gojjam — The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the women of West Gojjam between 15-49 years by measuring hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), C-reactive protocol (CRP), alpha-1-acid glycoprotein (AGP), plasma Zn (PZn), plasma retinol and retinol binding protein (RBP), respectively.
  Groups: Women of West Gojjam
Other: Children of West Gojjam — The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the children of West Gojjam between the age of 6-59 months by measuring hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), C-reactive protocol (CRP), alpha-1-acid glycoprotein (AGP), plasma Zn (PZn), plasma retinol and retinol binding protein (RBP), respectively.
  Groups: Children of West Gojjam
Other: Women of Kamashi — The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the women of Kamashi between 15-49 years by measuring hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), C-reactive protocol (CRP), alpha-1-acid glycoprotein (AGP), plasma Zn (PZn), plasma retinol and retinol binding protein (RBP), respectively.
  Groups: Women of Kamashi
Other: Children of Kamashi — The prevalence of Fe, Zn and vitamin A deficiency will be assessed in the children of Kamashi between 6-59 months by measuring hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), C-reactive protocol (CRP), alpha-1-acid glycoprotein (AGP), plasma Zn (PZn), plasma retinol and retinol binding protein (RBP), respectively.
  Groups: Children of Kamashi

SUMMARY:
To conduct a sub-regional micronutrient survey (SRMNS) assessing the prevalence of vitamin A, Zn, and Fe status in the country

DETAILED DESCRIPTION:
Background: In Ethiopia, biofortified staple crops, such as high vitamin A maize, high zinc (Zn) maize, high Zn wheat and high iron (Fe) common bean could have a beneficial impact on micronutrient status, as the regular varieties of these crops are eaten in significant amounts in some of the administrative regions. It is however, unknown in which region people would most benefit as data on vitamin A, Zn and Fe status in the different regions is too limited to efficiently target specific biofortification approaches.

Objective: The overall objective of the project is to generate data to target and tailor bio fortification approaches in Ethiopia. Therefore, it is planned to conduct a sub-regional micronutrient surveys (SRMNS) assessing the prevalence of vitamin A, Zn, and Fe status in the country.

Study design: The sub regional micronutrient survey (SRMNS) will have a cross-sectional design with one measuring point.

Study population: The SRMNS will be conducted in 600 children < 5 years of age and 600 women of reproductive age (18-45 years) living in the regions of Kamashi in Benishangul Gumuz, West Gojjam in Amhara, and Goma Gofa in Southern Nations, Nationalities and People's Regions (SNNP).

Main study parameters/endpoints: The prevalence of Fe, Zn and vitamin A deficiency will be assessed by measuring hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), C-reactive protocol (CRP), alpha-1-acid glycoprotein (AGP), plasma Zn (PZn), plasma retinol and retinol binding protein (RBP), respectively.

Significance: The study will generate important data on the vitamin A, Zn and Fe status of children and women for sub-regions in Ethiopia. Such sub-regional data will be more specific than common survey data and therefore be helpful to target bio fortification and identify the populations in Ethiopia who will benefit most from high nutrient crops.

ELIGIBILITY:
Inclusion Criteria:

* 5-59 months of age for children
* 15-49 years for women of reproductive age.
* The informed consent form has been read and signed by the caregiver (or has been read out to the caregiver in case of illiteracy)

Exclusion Criteria:

* Severely wasted and underweight children (weight for height and weight for age Z score < -3, respectively)
* Chronic or acute illness or other conditions that in the opinion of the Principle Investigator (PI) or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participants taking part in other studies requiring the drawing of blood
* Long-term medication (except contraceptives for women of reproductive age)
* Any severe metabolic, gastrointestinal kidney or chronic disease such as diabetes, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement or examination of study doctor). Health records to be checked for the same.
* Blood losses (surgery, accident), donations or transfusions during the past 4 months before study start.

Ages: 5 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — For the Children, both male and female are included. For adults, only women between ages of 15 and 49 are included.
Study Population: households that have a woman of reproductive age (15-49 yrs) and children between 5- 59 months of age will be chosen to be a part of the study
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Anaemia | March 2018
  Prevalence of iron deficiency with or without anemia
Prevalence of Zinc deficiency | March 2018
  Based on plasma Zinc concentration
Prevalence of Vitamin A deficiency | March 2018
  Measuring Vitamin A biomarkers

SECONDARY OUTCOMES:
Inflammation biomarkers | March 2018
  C reactive protein (CRP)
Anthropometric measurement - Height | March 2018
  height in cm
Anthropometric measurement - Weight | March 2018
  weight in Kg
Inflammation Biomarker | March 2018
  Alpha 1-acid glycoprotein (AGP)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, PhD, Principal Investigator — Professor and Head, Human Nutrition, Swiss Federal Institute of Technology (ETH) Zurich, Switzerland; Kaleab Baye, PhD, Principal Investigator — Assistant Professor and Head, Center for Food Science and Nutrition, Addis Ababa Univeristy, Ethiopia
Locations (2):
- Center for Food Science and Nutrition, Addis Ababa University, Addis Ababa, Ethiopia
- Swiss Federal Institute of Technology (ETH), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No